CLINICAL TRIAL: NCT07195825
Title: A Single-arm, Open-label, Single-dose Clinical Study to Evaluate the Safety and Tolerability of BBM-P002 for Stereotactic Bilateral Putamen Injection in the Treatment of Idiopathic Parkinson's Disease
Brief Title: A Clinical Study to Evaluate the Safety, and Tolerability of BBM-P002 in the Treatment of Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Xinzhi BioMed Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBM003-CLN001
Record Dates: First submitted 2025-09-10; First posted 2025-09-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: PD
Keywords: PD; gene therapy; Adeno-Associated Virus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm of BBM-P002 (Experimental): Single-dose treatment
  Interventions: Genetic: Injecting BBM-P002 into the bilateral putamen

INTERVENTIONS:
Genetic: Injecting BBM-P002 into the bilateral putamen — BBM-P002 is an AAV-based gene therapy that delivers a therapeutic gene cassette into putamen for the treatment of Parkinson's Disease

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of BBM-P002 for stereotactic injection to treat participants with idiopathic Parkinson's Disease (PD) during the dose-limiting toxicity (DLT) observation period.

DETAILED DESCRIPTION:
This is a single-arm, open-label study to evaluate the safety, tolerability, efficacy, pharmacokinetic, pharmacodynamic, and immune response of BBM-P002 within 52 weeks after into the bilateral putamen in Parkinson's disease, as well as the long-term safety and efficacy of BBM-P002 for up to 5 years post injection.

BBM-P002 is an AAV-based gene therapy that delivers a therapeutic gene cassette into putamen for the treatment of Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a diagnosis of Parkinson's disease for ≥ 5 years.
2. The Hoehn-Yahr staging meets the requirements during the OFF periods.
3. The MDS-UPDRS Part III score met the requirements during the OFF periods. the levodopa challenge test was positive
4. During the screening period, participants were required to take the same stable dose of dopamine-releasing drugs (such as levodopa) regularly
5. The participants agreed to postpone the neurosurgical procedures related to the indication treatment during the main study phase
6. The participants agreed not to participate in any other therapeutic intervention studies during the trial period
7. The participants agreed not to receive the vaccine during the main study phase
8. From the screening period until at least 52 weeks after dosing, use a reliable contraceptive method
9. The participants had good compliance and were able to undergo regular follow-ups. During the follow-up period, they were able to accurately complete the diary cards. Family members, guardians or caregivers could assist the subjects in filling out the diary cards
10. Voluntarilyvoluntarily participated in the study and signed the informed consent form

Exclusion Criteria:

1. Atypical or secondary Parkinsonism
2. Have contraindications for surgery or have previously undergone brain surgery
3. The participants has an abnormal brain MRI suggestive of brain pathology other than Parkinson's disease
4. Those with severe cognitive impairments
5. Those with severe depression or severe anxiety
6. Abnormal liver function
7. Abnormal coagulation function
8. Abnormalities in infectious disease screening
9. Currently undergoing antiviral treatment for hepatitis
10. Suffering from unstable or severe diseases in the cardiovascular, respiratory, digestive, nervous, hematological, immune and other systems
11. Suffering from malignant tumors or having a history of tumors
12. Previous history of severe allergies
13. Exclude those who have participated in other clinical trials within the past three months
14. Had received gene therapy during the screening period
15. Select those who have received stem cell treatment within the past 12 months
16. Exclude those who have used other investigational drugs within the past 4 weeks
17. During the screening period, if the individual had received live vaccines within the previous 2 months, or had a history of vaccination within the last 30 days, they would be excluded.
18. Having a history of alcohol dependence or drug addiction
19. Pregnant or lactating female participants
20. The situations that were determined by the investigator to be unsuitable for inclusion in the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-27 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events | Within 4 weeks
  To evaluate the rate of incidence of DLT events determined by the Safety Data Review Committee (SRC) in DLT observation period after injecting BBM-P002
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Within 4 weeks
  To evaluate the safety of BBM-P002 by AEs and SAEs.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Within 5 years
  To assess the long-term safety of BBM-P002 by AEs and SAEs
Changes in the titers of neutralizing antibodies and binding antibodies in the recombinant adenovirus capsid of blood | Within 5 years
  To assess changes in the titers of neutralizing antibodies and binding antibodies in the recombinant adenovirus capsid of blood after injecting BBM-P002
Changes in the results of the cranial MRI scan | Within 5 years
  To assess changes in the results of the cranial MRI scan after injecting BBM-P002
Changes from baseline in MDS - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) I/II/III/IV scores | Within 5 years
  The theoretical maximum total score of the MDS-UPDRS is 272 points. It comprehensively assesses the health status of Parkinson's disease patients by evaluating four major aspects: non-motor symptoms, daily activities, motor function, and motor complications. The higher the score, the more severe the condition
Changes from baseline in the Patient Global Impression of Improvement (PGI-I) scores | Within 5 years
  Choose a number from 1 to 7. The higher the number choosen, the worse the improvement.
Changes from baseline in the Clinical Global Impression of Improvement (CGI-I) scores | Within 5 years
  Choose a number from 1 to 7. The higher the number choosen, the worse the improvement.
Changes in the activity levels of gene expression products under18F-dopa PET scanning from baseline [striatum - occipital lobe average radioactivity count ratio] | Within 5 years
  To assess changes in the activity levels of gene expression products under18F-dopa PET scanning from baseline [striatum - occipital lobe average radioactivity count ratio] after injecting BBM-P002
Changes from baseline in daily levodopa dose or equivalent dose of levodopa | Within 5 years
  To assess changes from baseline in the levodopa dosage or levodopa equivalent dosage after injecting BBM-P002
Changes from baseline in the percentage at on time. | Within 5 years
  To assess changes from baseline in the percentage at on time after injecting BBM-P002

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, MD, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Jing Sun, MD, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No